CLINICAL TRIAL: NCT04145401
Title: Post Market Clinical Follow-Up Study for EVOLUTION® Revision Tibial System and EVOLUTION® Revision Constrained Condylar Knee (CCK) Femur With the EVOLUTION® CCK Tibial Insert
Brief Title: Post Market Clinical Follow-Up Study- EVOLUTION® Revision CCK
Status: Enrolling by invitation | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18K001
Record Dates: First submitted 2019-10-17; First posted 2019-10-30 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; traumatic arthritis; avascular necrosis; rheumatoid arthritis; correction of functional deformity; revision procedures
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Revision Knee implants — Primary knee arthroplasty or a revision knee that requires a revision procedure.

SUMMARY:
Sponsor is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its EVOLUTION® Revision CCK Tibia and EVOLUTION® Revision CCK Femur with EVOLUTION® CCK Tibial inserts. These type of studies are required by regulatory authorities for all devices that have been approved in Europe (EU) to evaluate the medium and long term clinical evidence. This study has been designed in accordance with MEDDEV2.12/2 rev 2 (European Medical Device Vigilance System) and ISO (International Organization for Standardization) 14155:2011 guidelines.

DETAILED DESCRIPTION:
The objectives of this study are:

1. To estimate the individual component survivorship of EVOLUTION® Revision Tibia, EVOLUTION® Revision CCK Femur, and EVOLUTION® CCK Tibial Insert.
2. To find out the cumulative incidence of component revision of each component in this combination.
3. To find out the functional outcome scores at early, midterm, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has been determined to undergo a revision knee arthroplasty that requires the study (EVOLUTION® Revision Tibial System and EVOLUTION® Revision CCK Femur with the EVOLUTION® CCK Tibial Insert)
2. Decision to perform the study index surgery with the required study components (EVOLUTION® Revision Tibial System and EVOLUTION® Revision CCK Femur with the EVOLUTION® CCK Tibial Insert) is pre-determined regardless of the research.
3. Previously implanted subjects must be enrolled within 3 years (+6 months) of their study index surgery
4. Willing and able to complete required study visits and assessments through the 10 year post-operative follow-up visit.

Bilateral subjects can have both TKAs enrolled in the study provided:

1. the specified combination of components (EVOLUTION® Revision Tibial System and EVOLUTION® Revision CCK Femur with the EVOLUTION® CCK Tibial Insert) were implanted in both
2. all other aspects of the Inclusion/Exclusion Criteria are satisfied
3. enrollment does not exceed the subject count specified
4. the subject agrees to a second Informed Consent document and data collection specific to the second TKA.

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation.
2. Has an overt infection at the time of implantation.
3. Has inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable.
4. Currently enrolled in another clinical investigation which would affect the endpoints of this protocol.
5. Has documented substance abuse issues.
6. Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study.
7. Currently incarcerated or has impending incarceration.
8. Has a medical condition, as judged by the Investigator, that would interfere with the subject's ability to comply with the requirements of the protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary TKA or Revision
  Single study group with either newly or previously implanted patients with EVOLUTION® Revision Tibia and EVOLUTION® Revision CCK Femur with the EVOLUTION® CCK Insert.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2033-05-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Individual component survivorship | 10 years post-operative
  Individual component survivorship for tibial base, femoral, and tibial insert at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient Reported Outcomes- Questionnaires | 10 years post-operative
  * functional scores for subjects, as assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS), out to 10 years follow-up
  * functional scores for subjects, as assessed by EuroQol-5D-5L (EQ-5D-5L) Scores, out to 10 years follow-up
  * subject satisfaction measures with their Total Knee Arthroplasty (TKA) procedure using the Forgotten Joint Score
  * subject satisfaction measures with their TKA procedure using the Satisfaction Survey
Incidence of component revision | 10 years post-operative
  the cumulative incidence of component revision at specified intervals will be determined out to 10 years follow-up
Radiolucencies | 10 years post-operative
  the presence, zone, and the size of radiolucencies surrounding implanted components will be determined
Adverse Events and Adverse Device Effects | 10 years post-operative
  characterization of adverse events and adverse device effects

CONTACTS AND LOCATIONS:
Locations (1):
- HCA Research Institute, OrthoONE at Swedish Medical Center, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No